CLINICAL TRIAL: NCT04836845
Title: Comparative Effects of Radial and Focused Extracorporeal Shock Wave Therapies on Calcaneal Spur: A Randomised Sham-controlled Trial
Brief Title: Comparation of Radial and Focused Extracorporeal Shock Waves in Calcaneal Spur: A Randomised Sham-controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Volkan Şah, Principal Investigator, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yuzuncu Yil University Van
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Calcaneal Spur
MeSH Terms: conditions — Heel Spur

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Focus extracorporeal shock wave therapy (Active Comparator)
  Interventions: Device: Focus extracorporeal shock wave therapy
- Radial extracorporeal shock wave therapy (Active Comparator)
  Interventions: Device: Radial extracorporeal shock wave therapy
- Sham extracorporeal shock wave therapy (Sham Comparator)
  Interventions: Device: Sham extracorporeal shock wave therapy

INTERVENTIONS:
Device: Focus extracorporeal shock wave therapy — Focus extracorporeal shock wave therapy, device: Electronica, Pagani, Italy
  Arms: Focus extracorporeal shock wave therapy
Device: Radial extracorporeal shock wave therapy — Radial extracorporeal shock wave therapy, device: Electronica, Pagani, Italy
  Arms: Radial extracorporeal shock wave therapy
Device: Sham extracorporeal shock wave therapy — Sham extracorporeal shock wave therapy, device: Electronica, Pagani, Italy
  Arms: Sham extracorporeal shock wave therapy

SUMMARY:
To date, focused and radial types of ESWT have been effectively used in calcaneal spur. However, studies directly addressing a comparison between radial and focused types of ESWT in calcaneal spur have not been done. Therefore, this study aims to evaluate comparative effects of radial and focused ESWT options on calcaneal spur.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of plantar calcaneal spur
* be aged ≥18 at the time of diagnosis
* be give informed consent

Exclusion Criteria:

* have not completed the assessment process.
* foot deformity
* psychological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 1 min.
  pain evaluation, higher scores mean a worse outcome.
American Orthopedic Foot and Ankle Score | 5 min.
  higher scores mean a better outcome.
FOOT FUNCTION INDEX | 7 min.
  higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyhmus Kaplan, Study Director — Yuzuncu Yil University
Locations (1):
- Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No